CLINICAL TRIAL: NCT01277536
Title: Explicit Assessment of Thromboembolic Risk and Prophylaxis for Medical Patients in Switzerland (ESTIMATE): Evaluation of a Prediction Rule
Brief Title: Explicit Assessment of Thromboembolic Risk and Prophylaxis for Medical Patients in Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Kantonsspital Baden (Other); University of Zurich (Other); Luzerner Kantonsspital (Other); Cantonal Hospital of St. Gallen (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Mathieu R NENDAZ, MD, University Hospital, Geneva
Other Study IDs: ESTIMATE
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hospitalization >24 hours

SUMMARY:
Until now, no risk assessment model informing about the need of thromboprophylaxis in patients admitted for an acute medical event has been validated.

The goal of this project is to indirectly validate a model developed in Geneva by a non -interventional study involving the collection of patient characteristics during the hospitalization and a 3-month follow-up. These data will allow for the determination of the patient's risk, according to the Geneva model, and its validity, according the actual thrombo-embolic events, corrected for the thromboprophylaxis received.

The project is multicentric in Switzerland (5-10 centers) and should involve about 1000 patients.

First amendment (may 2011) : we have obtained the IRB approval for collecting data from patients who die during their hospital stay and for whom informed consent is not be possible to obtain.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted (minimal stay >24 hours) to medical hospital wards
* Age ≥18 years
* Ability to give an informed consent, as informed by the physicians in charge of the patient

Exclusion Criteria:

* Patients admitted to non-medical hospital wards
* Patients with therapeutic anticoagulation at hospital admission
* Patients admitted for a disease requiring therapeutic anticoagulation (MTE or other)
* Patients unable to give an informed consent, as informed by the physicians in charge of the patient
* Patients without signed informed consent
* Patients already included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Several public hospitals of Switzerland, genral internal medicine divisions
Sampling Method: Non-Probability Sample
Enrollment: 1478 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
relationship between the combined rate of fatal and non-fatal symptomatic venous thromboembolism and bleeding events and the calculated risk score at 90 days after hospital admission | 90 days
  evaluation of the relationship between the combined rate of fatal and non-fatal symptomatic venous thromboembolism and bleeding events at 90 days after hospital admission on one hand, and the calculated risk score provided by the Geneva Risk Assessment Models (RAM) at hospital admission on the other hand

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu R Nendaz, Dr, Principal Investigator — General Internal Medicine Division, University Hospitals of Geneva
Locations (7):
- Switzerland (7):
  - Kantonsspital, Baden
  - University Hospitals, Bern
  - Cantonal Hospital, Fribourg
  - University Hospitals, Geneva
  - Kantonsspital, Lüzern
  - Cantonal Hospital, Sankt Gallen
  - University Hospital, Zurich

REFERENCES:
- [Background] Chopard P, Spirk D, Bounameaux H. Identifying acutely ill medical patients requiring thromboprophylaxis. J Thromb Haemost. 2006 Apr;4(4):915-6. doi: 10.1111/j.1538-7836.2006.01818.x. No abstract available. PMID 16634771
- [Result] Nendaz M, Spirk D, Kucher N, Aujesky D, Hayoz D, Beer JH, Husmann M, Frauchiger B, Korte W, Wuillemin WA, Jager K, Righini M, Bounameaux H. Multicentre validation of the Geneva Risk Score for hospitalised medical patients at risk of venous thromboembolism. Explicit ASsessment of Thromboembolic RIsk and Prophylaxis for Medical PATients in SwitzErland (ESTIMATE). Thromb Haemost. 2014 Mar 3;111(3):531-8. doi: 10.1160/TH13-05-0427. Epub 2013 Nov 14. PMID 24226257
- [Derived] Spirk D, Nendaz M, Aujesky D, Hayoz D, Beer JH, Husmann M, Frauchiger B, Korte W, Wuillemin WA, Righini M, Bounameaux H, Kucher N. Predictors of thromboprophylaxis in hospitalised medical patients. Explicit ASsessment of Thromboembolic RIsk and Prophylaxis for Medical PATients in SwitzErland (ESTIMATE). Thromb Haemost. 2015 May;113(5):1127-34. doi: 10.1160/TH14-06-0525. Epub 2015 Jan 22. PMID 25608607